CLINICAL TRIAL: NCT01589614
Title: A Phase 1, Randomised, Open Label, Two Sequence, Two Treatment, Two Way Crossover Study to Estimate the Steady-state Effect of Erythromycin on the Single Dose Pharmacokinetics of Ph-797804 in Healthy Subjects
Brief Title: A Study To Investigate The Effect Of Erythromycin On The Pharmacokinetics Of PH-797804
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A6631036
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Healthy
MeSH Terms: interventions — PH 797804; Erythromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PH-797804 6 mg (Experimental): Subjects will receive a single 6 mg dose in the fed state
  Interventions: Drug: PH-797804
- PH-797804 6 mg + erythromycin 800 mg (Experimental): Subjects will receive multiple 800 mg doses of erythromycin and a single 6 mg dose of PH-797804 in the fed state
  Interventions: Drug: PH-797804 + erythromycin

INTERVENTIONS:
Drug: PH-797804 — Tablet, 6mg, single
  Arms: PH-797804 6 mg
Drug: PH-797804 + erythromycin — PH-797804: tablet, 6mg, single erythromycin: tablet, 400 mg, multiple
  Arms: PH-797804 6 mg + erythromycin 800 mg

SUMMARY:
The purpose of this study is to investigate the effect of co-administration with erythromycin on the time course of PH-797804 concentration in the blood following dosing by oral immediate release tablet formulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects and/or healthy female subjects of non-child bearing potential between the ages of 21 and 55 years (inclusive). Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurements, 12-lead ECG and clinical laboratory tests.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight > 50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 21 drinks/week for males.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 0,1,2,3,4,6,8,12,24,48,72,96,120,144,168,192,216,240 hours post-dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0,1,2,3,4,6,8,12,24,48,72,96,120,144,168,192,216,240 hours post-dose
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0,1,2,3,4,6,8,12,24,48,72,96,120,144,168,192,216,240 hours post-dose
Plasma Decay Half-Life (t1/2) | 0,1,2,3,4,6,8,12,24,48,72,96,120,144,168,192,216,240 hours post-dose
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] | 0,1,2,3,4,6,8,12,24,48,72,96,120,144,168,192,216,240 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6631036&StudyName=A%20Study%20To%20Investigate%20The%20Effect%20Of%20Erythromycin%20On%20The%20Pharmacokinetics%20Of%20PH-797804%20